CLINICAL TRIAL: NCT07031817
Title: Validation of a Composite Medical Device Using a Blood Biomarker-based Algorithm and MDQ for the Diagnosis of Bipolar Disorder in Patients With a Characterized Depressive Episode in Primary Care
Brief Title: Validation of a Composite Medical Device Using a Blood Biomarker-based Algorithm and MDQ for the Diagnosis of Bipolar Disorder
Acronym: BIPOVITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: CH Béziers (Unknown); Centre Hospitalier Universitaire de Nīmes (Other); Assistance Publique Hopitaux De Marseille (Other); University Hospital, Toulouse (Other); Nantes University Hospital (Other); USSAP Carcassonne (Unknown); Ajaccio Hospital Center (Other); CH TOULON (Unknown); CH Thuir (Unknown); CH Montauban (Unknown); Centre de Ressources Biologiques de Montpellier (Unknown); Federation Regionale de Recherche en Psychiatrie et Sante Mentale Occitanie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0553
Record Dates: First submitted 2025-05-30; First posted 2025-06-22 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder (BD); Major Depressive Episode (MDE); Primary Care; Major Depression
Keywords: bipolar disorder; major depressive episode; primary care; composite medical device; blood biomarkers; mood depression questionnaire; diagnosis; composite diagnostic tool; in vitro diagnostic test; blood biomarker-based algorithm
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic Evaluation Arm (Experimental): Participants in this arm will undergo the full diagnostic procedure under investigation. This includes :
  * A blood sample collected for analysis by the investigational in vitro diagnostic device targeting biomarkers associated with bipolar disorder,
  * Completion of validated psychiatric questionnaires, including the Mood Disorder Questionnaire (MDQ), used as clinical reference standards,
  * Collection of sociodemographic and clinical data relevant to the psychiatric profile. This arm does not involve any therapeutic intervention. The objective is to evaluate the diagnostic concordance between the blood test and psychiatric screening tools.
  Interventions: Diagnostic Test: Venous blood sample for measuring blood biomarkers related to bipolar disorder; Other: Standardized psychiatric assessment tools

INTERVENTIONS:
Diagnostic Test: Venous blood sample for measuring blood biomarkers related to bipolar disorder — Participants will undergo a venous blood draw for analysis by an investigational composite medical device designed to aid in the diagnosis of bipolar disorder. The device analyzes specific circulating biomarkers hypothesized to differ between patients with bipolar disorder and those with unipolar depression.
Other: Standardized psychiatric assessment tools — Participants will complete validated psychiatric screening tools used as reference standards to evaluate bipolar disorder, including the Mood Disorder Questionnaire (MDQ). These tools will be used to compare their diagnostic output with that of the investigational blood test.

SUMMARY:
The goal of this interventional clinical trial is to assess the diagnostic performance of a composite diagnostic medical devise based on blood-based in vitro diagnostic device and Mood Disorder Questionnaire (MDQ) in identifying bipolar disorder among adult patients presenting with a current major depressive episode in primary care. The study will compare the results of the medical device diagnostic test to those of standardized psychiatric clinical evaluation, to evaluate its sensitivity, specificity, and overall clinical utility.

The main research questions are :

* Can the investigational medical device accurately distinguish bipolar disorder from unipolar depression ?
* How does its diagnostic accuracy compare with validated psychiatric questionnaires commonly used in clinical practice ?

Participants will :

* Provide a blood sample for biomarker analysis using the investigational diagnostic device.
* Complete a few validated psychiatric assessment tools (e.g., MDQ, MINI).
* Share sociodemographic and clinical data relevant to psychiatric evaluation.

DETAILED DESCRIPTION:
Introduction

Bipolar disorder (BD) is a chronic and disabling condition affecting between 1% to 2.5% of the population, corresponding to approximately 650,000 to 1,650,000 individuals in France. Onset typically occurs between the ages of 15 and 25, with symptoms persisting throughout life. Bipolar disorder ranks as the sixth leading cause of disability globally, according to the World Health Organization (WHO). Additionally, individuals with bipolar disorder face a reduced life expectancy of around 10 years compared with the general population. This increased mortality is partly attributed to suicide, as approximately 20% of untreated BD patients die by suicide. In addition, BD is associated with a high prevalence of comorbidities such as alcohol or substance use disorders, diabetes, dyslipidaemia, which significantly heighten the risk of developing other diseases, notably cardiovascular pathologies. Risky behaviors, including impulsive spending, substance use, and unsafe sexual practices, further contribute to the functional impairments experienced by those with bipolar disorder. Clinically, bipolar disorder is characterized by alternating episodes of depression and mania or hypomania. While mania and hypomania are hallmark features of bipolar disorder, depressive episodes are more frequent and often serve as the initial clinical manifestation. This overlap with Major Depressive Disorder presents diagnostic challenges, particularly since patients often seek treatment during depressive phases, usually from general practitioners.

Current diagnostic approaches for bipolar disorder rely heavily on clinical assessment, necessitating detailed knowledge of mood disorders and extensive patient interviews-both of which are often impractical in primary care settings. Consequently, many bipolar disorder patients are misdiagnosed with major depressive disorder and receive inappropriate treatment with antidepressants, which can exacerbate the condition. Studies indicate that the prevalence of undiagnosed bipolar disorder in patients treated with antidepressants ranges around 10% in primary care to 16%-47% in psychiatric settings. In this context, the average diagnostic delay of bipolar disorder is 8 years in France. Early diagnosis and treatment could significantly improve the outcomes for bipolar disorder patients.

Self-administered tools such as the Mood Disorder Questionnaire (MDQ) offer potential solutions to improve bipolar disorder screening. The MDQ evaluates symptoms of mania or hypomania through a structured questionnaire divided into three sections: (1) assessment of 13 symptoms related to mania/hypomania, (2) evaluation of symptom temporality, and (3) determination of symptom impact on daily life. Despite its simplicity and utility, the MDQ has notable limitations, including low sensitivity (43%) and high specificity (95%), which restricts its standalone diagnostic reliability in primary care settings.

In this context, the development of an in vitro diagnostic test based on blood biomarkers, enabling differential diagnosis between bipolar disorder and major depressive disorder in patients with major depressive episode, represents a critical advancement. Recent research underscored the potential utility of biomarkers to complement clinical evaluations and enhance diagnostic accuracy. A predictive model was developed incorporating routinely measured blood-based biomarkers, such as eosinophil counts, prolactin levels, total cholesterol (TC), and low-density lipoprotein (LDL) cholesterol, to differentiate bipolar disorder from major depressive disorder. Their nomogram demonstrated robust discriminatory power with an area under the curve (AUC) of 0.858, highlighting the promise of biomarker-based diagnostics. Another notable development in this area is the Edit-B® test, which utilizes RNA editing markers and was introduced in France in 2024. However, this test has faced regulatory challenges, emphasizing the need of alternative diagnostic solutions.

Building on these advancements, the principal investigator and collaborators have developed a novel diagnostic algorithm combining biomarker analysis with the MDQ. Preliminary data suggest that this composite tool can enhance diagnostic precision, particularly in primary care settings where traditional clinical assessments are constrained. The proposed algorithm integrates the strengths of the biomarker-based approach, notably its high sensitivity, with the MDQ's specificity, aiming to achieve a sensitivity exceeding 85% and a specificity above 80%.

This research seeks to validate the efficacy of this composite diagnostic tool, hypothesizing that its implementation will significantly improve bipolar disorder screening and diagnosis in primary care. By leveraging biomarker insights and patient-reported data, the study aims to reduce diagnostic delays, optimize treatment strategies, and ultimately improve outcomes for individuals with bipolar disorder. The results of this study have the potential to bridge the gap between research and clinical practice, offering a scalable and accessible diagnostic tool for psychiatric disorders.

This is a multicenter, prospective, with no comparator group interventional clinical trial aiming to evaluate the diagnostic performance of a blood-based medical device for the detection of bipolar disorder in adult patients presenting with a current major depressive episode in primary care. The study will be conducted in the psychiatry departments of the different hospitals in the project. Participants will be recruited in primary care settings during a consultation for a depressive episode. All eligible participants will provide written informed consent.

Objectives

The primary aim of this study is to assess the diagnostic performance of a composite medical device that combines a blood biomarker-based algorithm and the MDQ for diagnosing bipolar disorder in patients presenting with a major depressive episode in primary care settings. Specifically, the focus is on determining the sensitivity and specificity of this composite medical device.

Several secondary objectives will be explored in this study. First, the area under the curve, negative predictive value (NPV), and positive predictive value (PPV) of the composite medical device will be determined for diagnosing bipolar disorder in patients with major depressive episode in primary care. Additionally, the characteristics of false negatives (FN) and false positives (FP), identified by the composite medical device, will be described. These characteristics will include demographic factors (age, sex, BMI), depression severity, biological markers of inflammation, clinical and biological variables collected during the study, comorbid addictive conditions, and psychotropic treatments.

Another key secondary objective is to assess the composite medical device's ability to predict the onset of hypomanic symptoms at 8 weeks and the improvement of depressive symptoms at 8 weeks. All these objectives will be revisited by taking the re-evaluated diagnosis at 8 weeks as a reference, which will also consider the occurrence of manic or hypomanic symptoms.

The study will also compare the diagnostic performance of the composite medical device with the diagnosis proposed by the general practitioner general practitioner. Furthermore, the variability in biomarker measurements across operators, methods, and sites will be measured, as well as the acceptability of the composite medical device among both patients and general practitioners.

The medico-economic impact of the composite medical device, if used to diagnose bipolar disorder in primary care, will also be evaluated, considering its sensitivity, specificity, and overall acceptability. Lastly, the study will seek to identify which biomarkers, either previously described in the literature or routinely measured in blood tests, could further enhance the performance of the composite medical device.

Interventions and study timeline

The first visit will be a pre-screening visit (V1). The pre-screening will be carried out by a general practitioner in their office during routine care. At the end of this pre-screening, and with the patient's consent, the general practitioner at each recruitment center will send the patient's contact information to the designated principal investigator's team. The principal investigator's team will then contact the potential participant by phone to schedule the screening visit.

The second visit will be a screening visit (V2). It will be conducted through a telephone interview. The investigator team will provide the patient with all relevant information about the study, including its objectives, benefits, risks, and procedures. The patient will be informed of the relevant legal provisions and their rights.

The third visit (V3) will be the inclusion visit. It will take place at one of the participating study centers, and at least 12 hours after the V2 visit to provide the patient with sufficient time to decide whether or not to participate in the study, without unduly delaying the specialized consultation and subsequent therapeutic guidance. A maximum delay of 7 days between patient selection and inclusion will also be respected. At the start of this visit, patients will be asked to sign the informed consent form for participation in the study. The patient will be evaluated by one of the investigators or a member of their team using standardized tools, self-assessment questionnaires (including MDQ, HCL-32, QIDS), and hetero-questionnaires (including MINI, MADRS). An audio recording will be made during the MINI administration. An evaluation of the test's acceptability will be carried out using a Likert scale.

The fourth visit (V4) will be the visit during which a blood sample will be taken, between 7:00 AM and 11:00 AM, with the patient required to fast. This visit will take place either on the same day or within 3 days at most after the V3 visit. The collection will include two 2.5 mL Paxgene® tube for whole-blood RNA (ribonucleic acid), two 6 mL dry tube for serum, two 4 mL heparinized tube one for native DNA and one for plasma preparation and a 6 mL EDTA tube for complete blood count (retained for 15 years). These samples will be anonymised and sent to the Biological Resource Centre at Montpellier University Hospital. During V4 or immediately after V4, the general practitioner will be interviewed by the investigation team, either in person, via videoconference, or by email (secure medical messaging) regarding their diagnostic opinion (likelihood of bipolar disorder according to them on the Likert scale) and their view on the acceptability of the test. At the end of V4, the patient will be referred to their general practitioner or to any appropriate healthcare facility based on the diagnosis and the severity of the symptoms, with the patient's consent. A written or verbal care recommendation will be provided to the patient and their general practitioner, considering the evaluations carried out during V3.

The 5th visit (V5) will be a follow-up visit. It will take place between 7 and 9 weeks after V4 and will be conducted via telephone interview or teleconsultation. The visits will be conducted by the investigation team from the CHU of Montpellier or the centre where the inclusion took place, depending on team availability. The patient will be assessed by one of the investigators using standardized tools, self-questionnaires (inlcusingincluding the MDQ) completed online or in writing, and hetero-questionnaires. The investigator will document the treatment administered to the patient and their care path since V3 and determine how the depressive symptoms have evolved and whether hypomanic symptoms have appeared since V3. Following this interview, the investigator will make a new diagnosis, confirming or modifying the one made at V3.

Biological Sample Collection

Biological samples will be collected during the inclusion visit at each of the participating study centers and then temporarily stored in a freezer at -20°C.

Every 3 months, the biological samples will be shipped in a package containing dry ice to the CRB (Centre de Ressources Biologiques) in Montpellier, where it will be stored at -80°C. For biomarker measurements in serum, tubes containing 500 µl of serum (1 tube per patient) will be transported to the Institute of Molecular and Cellular Pharmacology, under the responsibility of Professor Nicolas Glaichenhaus before being used for biomarker measurement.

For the biomarker measurements necessary for the use of the composite medical device (DM), serum samples will be analysed using the V-PLEX® (Mesoscale Discovery) and Olink Flex® (Olink) platforms, following the protocols described by the manufacturers. Additional analyses on other platforms will also be carried out to address the secondary objectives, in the laboratory of Professor Lehman in Montpellier, Professor Glaichenhaus in Valbonne, Dr. Lutz in Strasbourg, or any other public or private research facility capable of meeting the study's objectives.

The collection of biological samples will be created and stored in compliance with regulations. It will be declared to the relevant regulatory authorities. The samples will be stored at -80°C at the CRB of the CHU of Montpellier for 12 years. A participant in the study may refuse for their biological samples to be stored in this collection.

The biological samples may be used to explore new blood biomarkers for bipolar disorder in patients with a mood disorder in primary care settings, which could lead to the creation of new medical devices or the exploration of new pathophysiological hypotheses.

Data Management and Statistical Methods

The study data will be entered through an electronic case report form (e-CRF) on the Ennov Clinical (Clinsight) software, which allows for real-time data quality control. All this patient data comes from source documents which are the original documents from which the data will be added to the e-CRF. The investigator undertakes to allow direct access to the study source data during control, audit or inspection visits.

In the data analysis, a brief description of the studied population will be presented. For each diagnostic test, the investigators will estimate the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), as well as the area under the ROC (Receiver Operating Characteristic) curve and their associated 95% confidence intervals.

To address the primary objective, the parameters of interest (sensitivity and specificity) for the primary outcome measure (sequential criterion) will be estimated both pointwise and by the 95% confidence interval. For secondary objectives, paired data comparison tests will be used for the various outcome measures.

The grey zones will be estimated according to the method of Cannesson et al.

If the performance of the biomarker-based algorithm and the MDQ are known, those of a composite medical device combining the two are difficult to predict, depending on whether the two tests are used in parallel or sequentially. To identify the most effective, the investigators will combine the biomarker-based algorithm and MDQ in four different ways :

* Parallel analysis using the biomarker-based algorithm and MDQ : Patients with the composite medical device (MD) will be those who are positive on both tests.
* Parallel analysis using the biomarker-based algorithm and MDQ : Positive patients with the composite MD will be those who are positive on at least one of the two tests.
* Sequential analysis using the biomarker-based algorithm and MDQ : Positive patients with the composite MD will be those, among those positive on the biomarker-based algorithm, who are positive on the MDQ.
* Sequential analysis using the biomarker-based algorithm and MDQ : Positive patients with the composite MD will be those, among those positive on the MDQ, who are positive on the biomarker-based algorithm.

The chosen composite MD will be the one that provides the best sensitivity and specificity, or the highest Youden index in the absence of an ordered relationship. The search for factors associated with misclassification errors will be done using multivariate analysis with logistic regression. Variables with a p-value <0.20 in univariate analysis will be included in the multivariate model. A forward selection procedure will then be used to obtain a final model.

A new composite score for the medical device will be determined through logistic regression. An individual score will be established for each patient using the coefficients from the multivariate logistic regression. Sensitivity, specificity, and predictive values will be calculated. The score's ability to predict patient status will be estimated by the AUC of the ROC curve and its associated 95% confidence interval. Various thresholds will be identified via the ROC curve based on the Youden index.

The variability in biomarker measurements according to the operator, laboratory, or platform usage will be assessed through the Intraclass Correlation Coefficient (ICC) calculations and the Bland-Altman graphical method. All tests will be two-tailed with an alpha risk set at 5%. A false discovery rate (FDR) penalty will be considered for the analysis of secondary criteria. For quality control purposes, diagnostic interviews will be re-listened to by an expert team, and the concordance between the diagnosis established by the investigator and the experts will be analysed by calculating Cohen's kappa index.

It will have two interim analyses, one after the inclusion of 200 patients and the other after the inclusion of 400 patients. During these two interim analyses, the prevalence of TB in the cohort of already included patients will be measured, as well as the sensitivity, specificity, PPV, NPV, and AUC of the composite MD using the diagnosis established at V3 as the reference.

The variability of biomarker measurements will be performed at each interim analysis. Biomarkers will be measured in parallel and independently in two different laboratories, specifically in the laboratories of Nicolas Glaichenhaus (CNRS) and Sylvain Lehmann (CHU of Montpellier).

ELIGIBILITY:
Inclusion Criteria :

* Cis man, cis woman, trans man, trans woman or non-binary,
* Aged 18 to 65 years old,
* Meets the DSM-5 criteria for the diagnosis of moderate to severe EDC and is eligible for antidepressant treatment.

Non-Inclusion Criteria :

* Patients under guardianship or trusteeship,
* Patients with schizophrenia according to DSM-5 criteria,
* Patients who have received psychotropic treatment in the 5 days prior to inclusion (or 21 days for fluoxetine or aripiprazole), with the exception of benzodiazepines and hydroxyzine at the doses and in compliance with the indications of the Marketing Authorisations,
* Patients with an unstable physiological state or a serious and symptomatic medical condition in the opinion of the investigator,
* Pregnant or breast-feeding patients,
* Patients with a known autoimmune disease, in particular Crohn's disease or thyroiditis, or any other pathology which could, in the opinion of the investigator, modify the blood concentration of immune biomarkers,
* Patients unable to give informed consent to participate in the study or who cannot be given informed information,
* Patients not covered by a social security scheme,
* Patients participating in another interventional study on the day of inclusion,
* Patients under court protection,
* Patients vaccinated less than 30 days ago,
* Patients with difficulties reading, understanding or speaking French.

Exclusion Criteria :

* Participants will have the right to withdraw their consent at any time for any reason whatsoever without any prejudice to them,
* The investigator may prematurely exclude a subject from the study, in agreement with the sponsor, if the subject presents one or more exclusion criteria,
* Diagnosis of schizophrenia during follow-up or any other diagnosis that would lead to a change in the initial EDC diagnosis,
* Any condition or situation which, in the opinion of the investigator, would be incompatible with the continuation of the study or which would lead to a bias in the management of the data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the composite medical device, using the full clinical evaluation as a reference | Through study completion, an 8 weeks follow-up for each patient
  To assess the sensitivity and specificity of a composite diagnostic device using a biomarker-based algorithm (IL-6, IL-10, IL-15, IL-27, CXCL10), combined with clinical data (age, depression severity via QIDS, psychotropic treatment), to identify bipolar disorder in primary care patients with a depressive episode. The algorithm, developed by the investigators, will be implemented in the eCRF and classify patients as bipolar, non-bipolar, or in a grey zone. The reference diagnosis will be established by an expert psychiatrist using the MINI interview and a full clinical evaluation, including medical history and patient records, following standardized procedures for optimal diagnostic accuracy.

SECONDARY OUTCOMES:
Area under the curve | Through study completion, an 8 weeks follow-up for each patient
  To determine the area under the curve (AUC) of the composite medical device for the diagnosis of bipolar disorder in patients presenting with a characterised depressive episode in primary care with a clinical assessment by an expert psychiatrist as reference.
Negative predictive value | Through study completion, an 8 weeks follow-up for each patient
  To determine the negative predictive value (NPV) of the composite medical device for the diagnosis of bipolar disorder in patients presenting with a characterised depressive episode in primary care with a clinical assessment by an expert psychiatrist as reference.
Positive predictive value | Through study completion, an 8 weeks follow-up for each patient
  To determine the positive predictive value (PPV) of the composite medical device for the diagnosis of bipolar disorder in patients presenting with a characterised depressive episode in primary care with a clinical assessment by an expert psychiatrist as reference.
Occurence of hypomanic symptoms | From inclusion to the last visit at 7/9 weeks later
  The occurrence of hypomanic symptoms will be determined by comparing the patient's responses to the MDQ at visit n°3 and visit n°5. Any positive response at visit n°5 to a question to which the response was negative at visit n°3 will indicate the occurrence of hypomanic symptoms between visit n°3 and visit n°5; if the number of hypomanic symptoms is greater at visit n°5 than at visit n°3, the patient will be classified in the 'new hypomanic symptoms' group.
Improvement in depression according to the MADRS scale | From inclusion to the last visit at 7/9 weeks later
  Improvement in depression will be defined as a reduction in symptomatology of at least 50% of the score on the MADRS between visit n°3 and visit n°5.
  Depressive symptoms are measured using the MADRS scale ; this scale corresponds to lists of symptoms whose presence and intensity are assessed by the patient or clinician. From 0 (No symtoms of depression) to 6 (Highest degree of symptoms). This allows an overall score to be calculated by adding up the scores for each item, with a higher score corresponding to greater intensity of depression. This scale is commonly used in research and clinical practice.
Improvement in depression according to the QIDS self-assessment questionnaire | From inclusion to the last visit at 7/9 weeks later
  Improvement in depression will be defined as a reduction in symptomatology of at least 50% of the score on the QIDS self-assessment questionnaire, between visit n°3 and visit n°5.
  Depressive symptoms are measured using the QIDS ; this questionnaire corresponds to lists of symptoms whose presence and intensity are assessed by the patient or clinician. This allows an overall score to be calculated by adding up the scores for each item, with a higher score corresponding to greater intensity of depression. This questionnaire is commonly used in research and clinical practice.
Improvement in depression according to the Patient Health Questionnaire (PHQ-9) self-assessment questionnaire | From inclusion to the last visit at 7/9 weeks later
  Improvement in depression will be defined as a reduction in symptomatology of at least 50% of the score on the PHQ-9, between visit n°3 and visit n°5.
  Depressive symptoms are measured using the PHQ-9 self-assessment questionnaire ; this questionnaire corresponds to lists of symptoms whose presence and intensity are assessed by the patient or clinician. This allows an overall score to be calculated by adding up the scores for each item, with a higher score corresponding to greater intensity of depression. This questionnaire is commonly used in research and clinical practice. The questionnaire is composed of 9 items : the minimum score is 0 and the maximum score is 3 for each item leading to a minimum total of 0 and maximum of 27.
Diagnosis of bipolar disorder | At the last visit between 7 and 9 weeks after inclusion
  The diagnosis of bipolar disorder at visit n°5 will be assessed in the same way as for the main objective.
Inter-operator variability in the measurement of biomarkers of bipolar disorder | Through study completion, an 8 weeks follow-up for each patient
  Measure inter-operator variability in the measurement of biomarkers used in composite medical device with all measurements from all the laboratories and measurement platforms used. It will be assessed through interclass correlation coefficient calculations and the Bland-Altman graphical method.
Inter-method variability in the measurement of biomarkers of bipolar disorder | Through study completion, an 8 weeks follow-up for each patient
  Measure inter-method variability in the measurement of biomarkers used in composite medical device with all measurements from all the laboratories and measurement platforms used. It will be assessed through interclass correlation coefficient calculations and the Bland-Altman graphical method.
Inter-site variability in the measurement of biomarkers of bipolar disorder | Through study completion, an 8 weeks follow-up for each patient
  Inter-site variability in the measurement of biomarkers used in composite medical device with all measurements from all the laboratories and measurement platforms used. It will be assessed through interclass correlation coefficient calculations and the Bland-Altman graphical method.
Acceptability of the composite medical device | Through study completion, an 8 weeks follow-up for each patient
  Acceptability of the medical dispositive for patients and general practitioners on a Likert scale. From 1 (Unacceptable) to 7 (Totally Acceptable).
Likert scale for the diagnosis of bipolar disorder in primary care | Through study completion, an 8 weeks follow-up for each patient
  The diagnosis of bipolar disorder in primary care will be collected from the general practitioner on a Likert scale of 1 (totally unlikely) to 7 (very highly likely), describing the probability of bipolar disorder.
Assay of ASAT (Aspartate Aminotransferase) | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (Ul/L).
Assay of ALAT (Alanine Aminotransferase) | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (Ul/L).
Assay of Alkaline Phosphatase | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (Ul/L).
Assay of GGT (Gamma-Glutamyl Transferase) | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (Ul/L).
Assay of Lactate Dehydrogenase (LDH) | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (Ul/L).
Assay of Total Bilirubin | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (µmol/L).
Assay of Conjugated Bilirubin | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (µmol/L).
Assay of Unconjugated Bilirubin | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (µmol/L).
Assay of Uric Acid | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (µmol/L).
Assay of Creatinine | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (µmol/L).
Assay of Triglycerides | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (g/L).
Assay of Total Cholesterol | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (g/L).
Assay of HDL Cholesterol | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (g/L).
Assay of LDL Cholesterol | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (g/L).
Assay of Albumin | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (g/L).
Assay of Urea | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (mmol/L).
Assay of CRP (C-Reactive Protein) | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (mg/L).
Assay of Free Triiodothyronine (FT3) | Through study completion, an 8 weeks follow-up for each patient
  A panel of routinely measured blood biomarkers will be assessed. These biomarkers will be analyzed either individually or as part of multivariate models, depending on their relevance to diagnostic accuracy. Measurements will be performed using immunoassays (V-PLEX, Olink) or standard clinical chemistry platforms. Outcomes will be reported in their respective standard units (pmol/L).
Medico-economic impact of the composite medical device | Through study completion, an 8 weeks follow-up for each patient
  For the medico-economic analysis, the costs of care and sick leave before and after the diagnosis of bipolar disorder on the basis of the SNDS (Système Nationale des Données de Santé). This analysis will be carried out in the general population without matching between the SNDS database and the patients included. The database will be shared with the medico-economic unit in order to weight the analysis by age and sex, for example. This strategy is justified in order to be able to use real data to assess the possible medical and economic impact of the composite medical device before and after the diagnosis of bipolar disorder. This objective cannot be achieved by data matching, since patients will be diagnosed at the time of study participation.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France

REFERENCES:
- [Background] Cannesson M. The "grey zone" or how to avoid the binary constraint of decision-making. Can J Anaesth. 2015 Nov;62(11):1139-42. doi: 10.1007/s12630-015-0465-1. Epub 2015 Aug 22. No abstract available. PMID 26296301
- [Background] Favre S, Aubry JM, Gex-Fabry M, Ragama-Pardos E, McQuillan A, Bertschy G. [Translation and validation of a French version of the Young Mania Rating Scale (YMRS)]. Encephale. 2003 Nov-Dec;29(6):499-505. French. PMID 15029084
- [Background] Sachs GS. Strategies for improving treatment of bipolar disorder: integration of measurement and management. Acta Psychiatr Scand Suppl. 2004;(422):7-17. doi: 10.1111/j.1600-0447.2004.00409.x. PMID 15330934
- [Background] Iannuzzo RW, Jaeger J, Goldberg JF, Kafantaris V, Sublette ME. Development and reliability of the HAM-D/MADRS interview: an integrated depression symptom rating scale. Psychiatry Res. 2006 Nov 29;145(1):21-37. doi: 10.1016/j.psychres.2005.10.009. Epub 2006 Oct 16. PMID 17049379
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Wiriyakijja P, Porter S, Fedele S, Hodgson T, McMillan R, Shephard M, Ni Riordain R. Validation of the HADS and PSS-10 and a cross-sectional study of psychological status in patients with recurrent aphthous stomatitis. J Oral Pathol Med. 2020 Mar;49(3):260-270. doi: 10.1111/jop.12991. Epub 2020 Jan 22. PMID 31919894
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Paquette D, Laporte L, Bigras M, Zoccolillo M. [Validation of the French version of the CTQ and prevalence of the history of maltreatment]. Sante Ment Que. 2004 Spring;29(1):201-20. doi: 10.7202/008831ar. French. PMID 15470573
- [Background] Gift TE, Reimherr ML, Marchant BK, Steans TA, Reimherr FW. Wender Utah Rating Scale: Psychometrics, clinical utility and implications regarding the elements of ADHD. J Psychiatr Res. 2021 Mar;135:181-188. doi: 10.1016/j.jpsychires.2021.01.013. Epub 2021 Jan 14. PMID 33493947
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Bech P, Christensen EM, Vinberg M, Bech-Andersen G, Kessing LV. From items to syndromes in the Hypomania Checklist (HCL-32): psychometric validation and clinical validity analysis. J Affect Disord. 2011 Jul;132(1-2):48-54. doi: 10.1016/j.jad.2011.01.017. Epub 2011 Feb 23. PMID 21349588
- [Background] Hirschfeld RM, Williams JB, Spitzer RL, Calabrese JR, Flynn L, Keck PE Jr, Lewis L, McElroy SL, Post RM, Rapport DJ, Russell JM, Sachs GS, Zajecka J. Development and validation of a screening instrument for bipolar spectrum disorder: the Mood Disorder Questionnaire. Am J Psychiatry. 2000 Nov;157(11):1873-5. doi: 10.1176/appi.ajp.157.11.1873. PMID 11058490
- [Background] Martinuzzi E, Barbosa S, Courtet P, Olie E, Guillaume S, Ibrahim EC, Daoudlarian D, Davidovic L, Glaichenhaus N, Belzeaux R. Blood cytokines differentiate bipolar disorder and major depressive disorder during a major depressive episode: Initial discovery and independent sample replication. Brain Behav Immun Health. 2021 Mar 10;13:100232. doi: 10.1016/j.bbih.2021.100232. eCollection 2021 May. PMID 34589747
- [Background] Carvalho AF, Takwoingi Y, Sales PM, Soczynska JK, Kohler CA, Freitas TH, Quevedo J, Hyphantis TN, McIntyre RS, Vieta E. Screening for bipolar spectrum disorders: A comprehensive meta-analysis of accuracy studies. J Affect Disord. 2015 Feb 1;172:337-46. doi: 10.1016/j.jad.2014.10.024. Epub 2014 Oct 23. PMID 25451435
- [Background] Boschloo L, Nolen WA, Spijker AT, Hoencamp E, Kupka R, Penninx BW, Schoevers RA. The Mood Disorder Questionnaire (MDQ) for detecting (hypo)manic episodes: its validity and impact of recall bias. J Affect Disord. 2013 Oct;151(1):203-8. doi: 10.1016/j.jad.2013.05.078. Epub 2013 Jun 20. PMID 23790555
- [Background] Scott J, Graham A, Yung A, Morgan C, Bellivier F, Etain B. A systematic review and meta-analysis of delayed help-seeking, delayed diagnosis and duration of untreated illness in bipolar disorders. Acta Psychiatr Scand. 2022 Nov;146(5):389-405. doi: 10.1111/acps.13490. Epub 2022 Sep 22. PMID 36018259
- [Background] Morselli PL, Elgie R; GAMIAN-Europe. GAMIAN-Europe/BEAM survey I--global analysis of a patient questionnaire circulated to 3450 members of 12 European advocacy groups operating in the field of mood disorders. Bipolar Disord. 2003 Aug;5(4):265-78. doi: 10.1034/j.1399-5618.2003.00037.x. PMID 12895204
- [Background] Vieta E. Antidepressants in bipolar I disorder: never as monotherapy. Am J Psychiatry. 2014 Oct;171(10):1023-6. doi: 10.1176/appi.ajp.2014.14070826. No abstract available. PMID 25272338
- [Background] McIntyre RS, Berk M, Brietzke E, Goldstein BI, Lopez-Jaramillo C, Kessing LV, Malhi GS, Nierenberg AA, Rosenblat JD, Majeed A, Vieta E, Vinberg M, Young AH, Mansur RB. Bipolar disorders. Lancet. 2020 Dec 5;396(10265):1841-1856. doi: 10.1016/S0140-6736(20)31544-0. PMID 33278937
- [Background] Vieta E, Berk M, Schulze TG, Carvalho AF, Suppes T, Calabrese JR, Gao K, Miskowiak KW, Grande I. Bipolar disorders. Nat Rev Dis Primers. 2018 Mar 8;4:18008. doi: 10.1038/nrdp.2018.8. PMID 29516993
- [Background] Aghababaie-Babaki P, Malekpour MR, Mohammadi E, Saeedi Moghaddam S, Rashidi MM, Ghanbari A, Heidari-Foroozan M, Esfahani Z, Mohammadi Fateh S, Hajebi A, Haghshenas R, Foroutan Mehr E, Rezaei N, Larijani B, Farzadfar F. Global, regional, and national burden and quality of care index (QCI) of bipolar disorder: A systematic analysis of the Global Burden of Disease Study 1990 to 2019. Int J Soc Psychiatry. 2023 Dec;69(8):1958-1970. doi: 10.1177/00207640231182358. Epub 2023 Jun 23. PMID 37353952
- [Derived] Fongaro E, Purper-Ouakil D, Picot MC, Epstein C, Kerbage H. Evaluating the effectiveness of telehealth-delivered Child and Family Traumatic Stress Intervention (CFTSI) for children and adolescents following recent trauma: a multi-zite randomized controlled trial in France. BMC Psychol. 2025 Nov 12;13(1):1254. doi: 10.1186/s40359-025-03585-0. PMID 41225581